CLINICAL TRIAL: NCT00067561
Title: A Twelve-Week, Randomized, Double Blind, Placebo-Controlled, Parallel-Group Study to Assess the Safety and Efficacy of 0.5 mg QD, 1 mg QD and 1 mg BID of Alosetron in Female Subjects With Severe Diarrhea-predominant IBS Who Have Failed Conventional Therapy
Brief Title: Study Of Women With Severe Diarrhea-Predominant Irritable Bowel Syndrome Having Failed Conventional Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S3B30040
Record Dates: First submitted 2003-08-21; First posted 2003-08-25 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Irritable Colon; Irritable Bowel Syndrome (IBS)
Keywords: Dose-ranging; Diarrhea-Predominant Irritable Bowel Syndrome; d-IBS; IBS; Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — alosetron

INTERVENTIONS:
Drug: Alosetron

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of different doses of an investigational medication in women with severe diarrhea-predominant Irritable Bowel Syndrome (IBS) who have failed conventional therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with severe diarrhea-predominant Irritable Bowel Syndrome (IBS).
* Failed conventional therapy.
* Willing to make daily calls on a touch-tone telephone.

Exclusion criteria:

* History of or current chronic or severe constipation.
* Bloody diarrhea, abdominal pain with rectal bleeding.
* Thrombophlebitis.
* Abnormal thyroid stimulating hormone (TSH) value.
* Alcohol and/or substance abuse within past two years.
* Pregnant or lactating.
* History/treatment of malignancy within past five years.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 702 (Actual)
Dates: Start 2003-06; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Subject self assessment of improvement between treatment groups using the IBS Global Improvement Scale; comparison of safety and tolerability between treatment groups with respect to adverse events & laboratory abnormalities.

SECONDARY OUTCOMES:
Comparison of treatment groups with respect to subject relief of IBS pain & discomfort.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (153):
- United States (152):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Calera, Alabama
  - GSK Investigational Site, Tuscaloosa, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Fayetteville, Arkansas
  - GSK Investigational Site, Chula Vista, California
  - GSK Investigational Site, Fountain Valley, California
  - GSK Investigational Site, Garden Grove, California
  - GSK Investigational Site, Lancaster, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Rancho Cucamonga, California
  - GSK Investigational Site, Redlands, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, San Rafael, California
  - GSK Investigational Site, Santa Ana, California
  - GSK Investigational Site, Upland, California
  - GSK Investigational Site, Vista, California
  - GSK Investigational Site, Yuba City, California
  - GSK Investigational Site, Boulder, Colorado
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Englewood, Colorado
  - GSK Investigational Site, Wheat Ridge, Colorado
  - GSK Investigational Site, Manchester, Connecticut
  - GSK Investigational Site, Boca Raton, Florida
  - GSK Investigational Site, Boynton Beach, Florida
  - GSK Investigational Site, Coral Gables, Florida
  - GSK Investigational Site, Fort Myers, Florida
  - GSK Investigational Site, Hialeah, Florida
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Lake Worth, Florida
  - GSK Investigational Site, Longwood, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Naples, Florida
  - GSK Investigational Site, New Port Richey, Florida
  - GSK Investigational Site, Ocala, Florida
  - GSK Investigational Site, Panama City, Florida
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, Tallahassee, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Zephyrhills, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Austell, Georgia
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Martinez, Georgia
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Peoria, Illinois
  - GSK Investigational Site, Riverside, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, South Bend, Indiana
  - GSK Investigational Site, Overland Park, Kansas
  - GSK Investigational Site, Bowling Green, Kentucky
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Madisonville, Kentucky
  - GSK Investigational Site, Davenport, Louisiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Laurel, Maryland
  - GSK Investigational Site, Silver Spring, Maryland
  - GSK Investigational Site, Towson, Maryland
  - GSK Investigational Site, Attleboro, Massachusetts
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Grand Rapids, Michigan
  - GSK Investigational Site, Oak Park, Michigan
  - GSK Investigational Site, Saint Joseph, Michigan
  - GSK Investigational Site, Warren, Michigan
  - GSK Investigational Site, Chaska, Minnesota
  - GSK Investigational Site, Saint Paul, Minnesota
  - GSK Investigational Site, Wentzville, Minnesota
  - GSK Investigational Site, Jackson, Mississippi
  - GSK Investigational Site, Jefferson City, Missouri
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Missoula, Montana
  - GSK Investigational Site, Lebanon, New Hampshire
  - GSK Investigational Site, Bloomfield, New Jersey
  - GSK Investigational Site, Egg Harbor, New Jersey
  - GSK Investigational Site, Ocean City, New Jersey
  - GSK Investigational Site, Vineland, New Jersey
  - GSK Investigational Site, West Caldwell, New Jersey
  - GSK Investigational Site, Farmington, New Mexico
  - GSK Investigational Site, Bay Shore, New York
  - GSK Investigational Site, Great Neck, New York
  - GSK Investigational Site, Merrick, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Stony Brook, New York
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, Asheville, North Carolina
  - GSK Investigational Site, Cary, North Carolina
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Fayetteville, North Carolina
  - GSK Investigational Site, Greenville, North Carolina
  - GSK Investigational Site, Hickory, North Carolina
  - GSK Investigational Site, High Point, North Carolina
  - GSK Investigational Site, Morehead City, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Bismarck, North Dakota
  - GSK Investigational Site, Akron, Ohio
  - GSK Investigational Site, Beavercreek, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Kettering, Ohio
  - GSK Investigational Site, Lyndhurst, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Altoona, Pennsylvania
  - GSK Investigational Site, Fleetwood, Pennsylvania
  - GSK Investigational Site, Hershey, Pennsylvania
  - GSK Investigational Site, Lancaster, Pennsylvania
  - GSK Investigational Site, Newtown, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Wyomissing, Pennsylvania
  - GSK Investigational Site, East Providence, Rhode Island
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Simpsonville, South Carolina
  - GSK Investigational Site, Bristol, Tennessee
  - GSK Investigational Site, Kingsport, Tennessee
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Murfreesboro, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Arlington, Texas
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Corpus Christi, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Humble, Texas
  - GSK Investigational Site, Irving, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Sugar Land, Texas
  - GSK Investigational Site, Tomball, Texas
  - GSK Investigational Site, Bountiful, Utah
  - GSK Investigational Site, Ogden, Utah
  - GSK Investigational Site, West Jordan, Utah
  - GSK Investigational Site, Alexandria, Virginia
  - GSK Investigational Site, Charlottesville, Virginia
  - GSK Investigational Site, Chesapeake, Virginia
  - GSK Investigational Site, Lacey, Washington
  - GSK Investigational Site, Spokane, Washington
  - GSK Investigational Site, Walla Walla, Washington
  - GSK Investigational Site, Wenatchee, Washington
  - GSK Investigational Site, Yakima, Washington
  - GSK Investigational Site, Milwaukee, Wisconsin
- GSK Investigational Site, Nedlands, Western Australia, Australia